CLINICAL TRIAL: NCT00000514
Title: Systolic Hypertension in the Elderly Program (SHEP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 33
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2005-01

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Disorders; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Cerebrovascular Disorders; Heart Diseases; Hypertension | interventions — Chlorthalidone; Atenolol; Reserpine

INTERVENTIONS:
Drug: chlorthalidone
Drug: atenolol
Drug: reserpine

SUMMARY:
The primary objective was to assess whether long-term administration of antihypertensive therapy to elderly subjects with isolated systolic hypertension reduced the combined incidence of fatal and non-fatal stroke. The secondary objectives were to evaluate: the effect of long-term antihypertensive therapy on mortality from any cause in elderly people with isolated systolic hypertension; possible adverse effects of chronic use of antihypertensive drug treatment in this population; the effect of therapy on indices of quality-of-life; the natural history of isolated systolic hypertension in the placebo population.

DETAILED DESCRIPTION:
BACKGROUND:

More than 3 million persons in the United States over the age of 60 have isolated systolic hypertension. They face an excess risk (2-3 fold) of stroke, other cardiovascular disease and death. Population-based data show that the prevalence rises from approximately 8 percent in the age group 60-69 years to approximately 20 percent over the age of 80. Based on available data, an annual stroke rate of 2.0 percent has been estimated in this population. The full-scale clinical trial followed a pilot study conducted from 1980 to 1983. Recruitment in the trial began in March 1985 and was finished in January 1988. Follow-up ended in February 1991. Data analysis continued through October 1996.

DESIGN NARRATIVE:

A randomized, double-blind trial in which 2,365 subjects were assigned to active treatment and 2,371 to placebo. For the active treatment group, a stepped-care regimen was used which included chlorthalidone 12.5 or 25 mg/day, and as needed, addition of atenolol 25 or 50 mg/day or reserpine, 0.05 or 0.10 mg/day. Treatment goal was to reduce systolic blood pressure by at least 20 mm Hg from baseline and to below 160 mm Hg with minimal amounts of study medication. The primary endpoint was the incidence of fatal and non-fatal stroke. Secondary endpoints were cardiovascular and coronary morbidity and mortality, all-cause mortality, and quality-of-life measures.

ELIGIBILITY:
Men and women, aged 60 or over, with isolated systolic hypertension.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1984-06; Study Completion 1996-10

CONTACTS AND LOCATIONS:
Overall Officials: C. Hawkins — University of Texas

REFERENCES:
- [Background] Hulley SB, Feigal D, Ireland C, Kuller LH, Smith WM. Systolic hypertension in the elderly program (SHEP). The first three months. J Am Geriatr Soc. 1986 Feb;34(2):101-5. doi: 10.1111/j.1532-5415.1986.tb05476.x. No abstract available. PMID 3511131
- [Background] Furberg CD, Cutler JA, Probstfield JL, et al: The Systolic Hypertension in the Elderly Program. Mild Hypertension: From Drug Trials to Practice, Raven Press, New York, 59-63, 1987.
- [Background] Rationale and design of a randomized clinical trial on prevention of stroke in isolated systolic hypertension. The Systolic Hypertension in the Elderly Program (SHEP) Cooperative Research Group. J Clin Epidemiol. 1988;41(12):1197-208. doi: 10.1016/0895-4356(88)90024-8. PMID 2905387
- [Background] Probstfield JL, Applegate WB, Curb JD, et al for the SHEP Cooperative Research Group: The Systolic Hypertension in the Elderly Program (SHEP): Rationale, Design, Recruitment, and Baseline Data. In: Omae T, Zanchetti A, (Eds.) How Should Elderly Hypertensive Patients Be Treated? Tokyo: Springer-Verlag, 135-142, 1989.
- [Background] Probstfield JL, Applegate WB, Borhani NO, Curb JD, Cutler JA, Davis BR, Furberg CD, Hawkins CM, Lakatos E, Page LB, et al. The Systolic Hypertension in the Elderly Program (SHEP): an intervention trial on isolated systolic hypertension. SHEP Cooperative Research Group. Clin Exp Hypertens A. 1989;11(5-6):973-89. doi: 10.3109/10641968909035386. PMID 2676266
- [Background] Schron EB, Davey JA, Jensen JM, Probstfield JL. The systolic hypertension in the elderly program. Implications for nursing practice and research. Prog Cardiovasc Nurs. 1989 Oct-Dec;4(4):138-45. PMID 2690065
- [Background] Pearson AC, Gudipati C, Nagelhout D, Sear J, Cohen JD, Labovitz AJ. Echocardiographic evaluation of cardiac structure and function in elderly subjects with isolated systolic hypertension. J Am Coll Cardiol. 1991 Feb;17(2):422-30. doi: 10.1016/s0735-1097(10)80109-3. PMID 1825095
- [Background] Prevention of stroke by antihypertensive drug treatment in older persons with isolated systolic hypertension. Final results of the Systolic Hypertension in the Elderly Program (SHEP). SHEP Cooperative Research Group. JAMA. 1991 Jun 26;265(24):3255-64. PMID 2046107
- [Background] Applegate WB, Davis BR, Black HR, Smith WM, Miller ST, Burlando AJ. Prevalence of postural hypotension at baseline in the Systolic Hypertension in the Elderly Program (SHEP) cohort. J Am Geriatr Soc. 1991 Nov;39(11):1057-64. doi: 10.1111/j.1532-5415.1991.tb02869.x. PMID 1753042
- [Background] Systolic Hypertension in the Elderly Program (SHEP). Baseline Characteristics of the Randomized Participants. Black HR, Curb JD, Pressel S, et al, Guest Editors.
- [Background] Borhani NO, Applegate WB, Cutler JA, Davis BR, Furberg CD, Lakatos E, Page L, Perry HM, Smith WM, Probstfield JL. Systolic Hypertension in the Elderly Program (SHEP). Part 1: Rationale and design. Hypertension. 1991 Mar;17(3 Suppl):II2-15. doi: 10.1161/01.hyp.17.3_suppl.ii2. No abstract available. PMID 1999373
- [Background] Petrovitch H, Byington R, Bailey G, Borhani P, Carmody S, Goodwin L, Harrington J, Johnson HA, Johnson P, Jones M, et al. Systolic Hypertension in the Elderly Program (SHEP). Part 2: Screening and recruitment. Hypertension. 1991 Mar;17(3 Suppl):II16-23. doi: 10.1161/01.hyp.17.3_suppl.ii16. No abstract available. PMID 1999371
- [Background] Vogt TM, Schron E, Pressel S, Wasserthiel-Smoller S, Eddleman EE, Miller S, Stamler J. Systolic Hypertension in the Elderly Program (SHEP). Part 3: Sociodemographic characteristics. Hypertension. 1991 Mar;17(3 Suppl):II24-34. doi: 10.1161/01.hyp.17.3_suppl.ii24. No abstract available. PMID 1999374
- [Background] Curb JD, Lee M, Jensen J, Applegate W. Systolic Hypertension in the Elderly Program (SHEP). Part 4: Baseline medical history findings. Hypertension. 1991 Mar;17(3 Suppl):II35-61. doi: 10.1161/01.hyp.17.3_suppl.ii35. No abstract available. PMID 1999375
- [Background] Labarthe DR, Blaufox MD, Smith WM, Lacy CR, Schnaper H, LaBaw F, Mascioli S, Davey J, Lakatos E. Systolic Hypertension in the Elderly Program (SHEP). Part 5: Baseline blood pressure and pulse rate measurements. Hypertension. 1991 Mar;17(3 Suppl):II62-76. doi: 10.1161/01.hyp.17.3_suppl.ii62. No abstract available. PMID 1999376
- [Background] Black HR, Unger D, Burlando A, Wright JC, Pressel SL, Allen R, McDonald RH, Surath H. Systolic Hypertension in the Elderly Program (SHEP). Part 6: Baseline physical examination findings. Hypertension. 1991 Mar;17(3 Suppl):II77-101. doi: 10.1161/01.hyp.17.3_suppl.ii77. No abstract available. PMID 1999377
- [Background] Hall WD, Davis BR, Frost P, Hoffmeier M, O'Brien JE, Pace S, Page L, Schneider KA, Stamler J. Systolic Hypertension in the Elderly Program (SHEP). Part 7: Baseline laboratory characteristics. Hypertension. 1991 Mar;17(3 Suppl):II102-22. doi: 10.1161/01.hyp.17.3_suppl.ii102. No abstract available. PMID 1999369
- [Background] Kostis JB, Prineas R, Curb JD, Lee M, Berkson D, Raines J, Frishman W, Francis CK, Sheffield T. Systolic Hypertension in the Elderly Program (SHEP). Part 8: Electrocardiographic characteristics. Hypertension. 1991 Mar;17(3 Suppl):II123-51. doi: 10.1161/01.hyp.17.3_suppl.ii123. No abstract available. PMID 1825649
- [Background] Weiler PG, Camel GH, Chiappini M, Greenlick MR, Hughes GH, Luhr JC, Moye LA, Mungas D, Perron M, Peters MH, et al. Systolic Hypertension of the Elderly Program (SHEP). Part 9: Behavioral characteristics. Hypertension. 1991 Mar;17(3 Suppl):II152-61. doi: 10.1161/01.hyp.17.3_suppl.ii152. No abstract available. PMID 1999370
- [Background] Implications of the systolic hypertension in the elderly program. The Systolic Hypertension in the Elderly Program Cooperative Research Group. Hypertension. 1993 Mar;21(3):335-43. PMID 8478043
- [Background] Davis BR, Wittes J, Pressel S, Berge KG, Hawkins CM, Lakatos E, Moye LA, Probstfield JL. Statistical considerations in monitoring the Systolic Hypertension in the Elderly Program (SHEP). Control Clin Trials. 1993 Oct;14(5):350-61. doi: 10.1016/0197-2456(93)90051-e. PMID 8222667
- [Background] Kostis JB, Allen R, Berkson DM, Curb JD, Davey J, Grimm RH, Hall WD, Lacy CR, Lee M, Miller S, et al. Correlates of ventricular ectopic activity in isolated systolic hypertension. SHEP Cooperative Research Group. Am Heart J. 1994 Jan;127(1):112-21. doi: 10.1016/0002-8703(94)90516-9. PMID 7506007
- [Background] Moye LA, Davis BR, Hawkins CM, Probstfield JL. Conclusions and implications of the systolic hypertension in the elderly program. Clin Exp Hypertens. 1993 Nov;15(6):911-24. doi: 10.3109/10641969309037081. PMID 8268898
- [Background] Frost PH, Davis BR, Burlando AJ, Curb JD, Guthrie GP Jr, Isaacsohn JL, Wassertheil-Smoller S, Wilson AC, Stamler J. Serum lipids and incidence of coronary heart disease. Findings from the Systolic Hypertension in the Elderly Program (SHEP). Circulation. 1996 Nov 15;94(10):2381-8. doi: 10.1161/01.cir.94.10.2381. PMID 8921777
- [Background] Curb JD, Pressel SL, Cutler JA, Savage PJ, Applegate WB, Black H, Camel G, Davis BR, Frost PH, Gonzalez N, Guthrie G, Oberman A, Rutan GH, Stamler J. Effect of diuretic-based antihypertensive treatment on cardiovascular disease risk in older diabetic patients with isolated systolic hypertension. Systolic Hypertension in the Elderly Program Cooperative Research Group. JAMA. 1996 Dec 18;276(23):1886-92. PMID 8968014
- [Background] Wassertheil-Smoller S, Applegate WB, Berge K, Chang CJ, Davis BR, Grimm R Jr, Kostis J, Pressel S, Schron E. Change in depression as a precursor of cardiovascular events. SHEP Cooperative Research Group (Systoloc Hypertension in the elderly). Arch Intern Med. 1996 Mar 11;156(5):553-61. PMID 8604962
- [Background] Frost PH, Davis BR, Burlando AJ, Curb JD, Guthrie GP, Isaacsohn JL, Wassertheil-Smoller S, Wilson AC, Stamler J. Coronary heart disease risk factors in men and women aged 60 years and older: findings from the Systolic Hypertension in the Elderly Program. Circulation. 1996 Jul 1;94(1):26-34. doi: 10.1161/01.cir.94.1.26. PMID 8964114
- [Background] Borhani NO. Risk management in stroke prevention: major clinical trials in hypertension. Health Rep. 1994;6(1):76-86. English, French. PMID 7919093
- [Background] Staessen JA, Amery A, Birkenhager W. Inverse association between baseline pressure and benefit from treatment in isolated systolic hypertension. Hypertension. 1994 Feb;23(2):269-70. doi: 10.1161/01.hyp.23.2.269. No abstract available. PMID 8307638
- [Background] Bearden D, Allman R, McDonald R, Miller S, Pressel S, Petrovitch H. Age, race, and gender variation in the utilization of coronary artery bypass surgery and angioplasty in SHEP. SHEP Cooperative Research Group. Systolic Hypertension in the Elderly Program. J Am Geriatr Soc. 1994 Nov;42(11):1143-9. doi: 10.1111/j.1532-5415.1994.tb06979.x. PMID 7963199
- [Background] Kostis JB, Lacy CR, Hall WD, Wilson AC, Borhani NO, Krieger SD, Cosgrove NM. The effect of chlorthalidone on ventricular ectopic activity in patients with isolated systolic hypertension. The SHEP Study Group. Am J Cardiol. 1994 Sep 1;74(5):464-7. doi: 10.1016/0002-9149(94)90904-0. PMID 7520210
- [Background] Applegate WB, Pressel S, Wittes J, Luhr J, Shekelle RB, Camel GH, Greenlick MR, Hadley E, Moye L, Perry HM Jr, et al. Impact of the treatment of isolated systolic hypertension on behavioral variables. Results from the systolic hypertension in the elderly program. Arch Intern Med. 1994 Oct 10;154(19):2154-60. PMID 7944835
- [Background] Hertert S, Bailey G, Cottinghan V, Carmody S, Egan D, Johnson P, Probstfield J. Community volunteers as recruitment staff in a clinical trial: the systolic hypertension in the elderly program (SHEP) experience. Control Clin Trials. 1996 Feb;17(1):23-32. doi: 10.1016/0197-2456(95)00074-7. PMID 8721799
- [Background] Kostis JB, Davis BR, Cutler J, Grimm RH Jr, Berge KG, Cohen JD, Lacy CR, Perry HM Jr, Blaufox MD, Wassertheil-Smoller S, Black HR, Schron E, Berkson DM, Curb JD, Smith WM, McDonald R, Applegate WB. Prevention of heart failure by antihypertensive drug treatment in older persons with isolated systolic hypertension. SHEP Cooperative Research Group. JAMA. 1997 Jul 16;278(3):212-6. PMID 9218667
- [Background] Applegate WB. Quality of life during antihypertensive treatment. Lessons from the Systolic Hypertension in the Elderly Program. Am J Hypertens. 1998 Mar;11(3 Pt 2):57S-61S. doi: 10.1016/s0895-7061(98)00012-0. No abstract available. PMID 9546039
- [Background] Davis BR, Vogt T, Frost PH, Burlando A, Cohen J, Wilson A, Brass LM, Frishman W, Price T, Stamler J. Risk factors for stroke and type of stroke in persons with isolated systolic hypertension. Systolic Hypertension in the Elderly Program Cooperative Research Group. Stroke. 1998 Jul;29(7):1333-40. doi: 10.1161/01.str.29.7.1333. PMID 9660383
- [Background] Pahor M, Shorr RI, Somes GW, Cushman WC, Ferrucci L, Bailey JE, Elam JT, Applegate WB. Diuretic-based treatment and cardiovascular events in patients with mild renal dysfunction enrolled in the systolic hypertension in the elderly program. Arch Intern Med. 1998 Jun 22;158(12):1340-5. doi: 10.1001/archinte.158.12.1340. PMID 9645829
- [Background] Cosgrove N, Borhani NO, Bailey G, Borhani P, Levin J, Hoffmeier M, Krieger S, Lovato LC, Petrovitch H, Vogt T, Wilson AC, Breeson V, Probstfield JL. Mass mailing and staff experience in a total recruitment program for a clinical trial: the SHEP experience. Systolic Hypertension in the Elderly Program. Cooperative Research Group. Control Clin Trials. 1999 Apr;20(2):133-48. doi: 10.1016/s0197-2456(98)00055-5. PMID 10227414
- [Background] Savage PJ, Pressel SL, Curb JD, Schron EB, Applegate WB, Black HR, Cohen J, Davis BR, Frost P, Smith W, Gonzalez N, Guthrie GP, Oberman A, Rutan G, Probstfield JL, Stamler J. Influence of long-term, low-dose, diuretic-based, antihypertensive therapy on glucose, lipid, uric acid, and potassium levels in older men and women with isolated systolic hypertension: The Systolic Hypertension in the Elderly Program. SHEP Cooperative Research Group. Arch Intern Med. 1998 Apr 13;158(7):741-51. doi: 10.1001/archinte.158.7.741. PMID 9554680
- [Background] Wittes J, Lakatos E, Black D, Geraci B, Davis B, Moye L, Probstfield J. Selecting screening criteria for clinical trials: an example from the Systolic Hypertension in the Elderly Program. Control Clin Trials. 1999 Apr;20(2):121-32. doi: 10.1016/s0197-2456(98)00047-6. PMID 10227413
- [Background] Perry HM Jr, Davis BR, Price TR, Applegate WB, Fields WS, Guralnik JM, Kuller L, Pressel S, Stamler J, Probstfield JL. Effect of treating isolated systolic hypertension on the risk of developing various types and subtypes of stroke: the Systolic Hypertension in the Elderly Program (SHEP). JAMA. 2000 Jul 26;284(4):465-71. doi: 10.1001/jama.284.4.465. PMID 10904510
- [Background] Wassertheil-Smoller S, Fann C, Allman RM, Black HR, Camel GH, Davis B, Masaki K, Pressel S, Prineas RJ, Stamler J, Vogt TM. Relation of low body mass to death and stroke in the systolic hypertension in the elderly program. The SHEP Cooperative Research Group. Arch Intern Med. 2000 Feb 28;160(4):494-500. doi: 10.1001/archinte.160.4.494. PMID 10695689
- [Background] Kostis JB, Lawrence-Nelson J, Ranjan R, Wilson AC, Kostis WJ, Lacy CR. Association of increased pulse pressure with the development of heart failure in SHEP. Systolic Hypertension in the Elderly (SHEP) Cooperative Research Group. Am J Hypertens. 2001 Aug;14(8 Pt 1):798-803. doi: 10.1016/s0895-7061(01)02044-1. PMID 11497197
- [Background] Kostis JB, Wilson AC, Freudenberger RS, Cosgrove NM, Pressel SL, Davis BR; SHEP Collaborative Research Group. Long-term effect of diuretic-based therapy on fatal outcomes in subjects with isolated systolic hypertension with and without diabetes. Am J Cardiol. 2005 Jan 1;95(1):29-35. doi: 10.1016/j.amjcard.2004.08.059. PMID 15619390
- [Background] Wittes J, Davis B, Berge K, Cohen JD, Grimm RH Jr, Hawkins CM, Kuller L. Systolic Hypertension of the Elderly Program (SHEP). Part 10: Analysis. Hypertension. 1991 Mar;17(3 Suppl):II162-7. doi: 10.1161/01.hyp.17.3_suppl.ii162. PMID 1999372
- [Background] Winker MA, Murphy MB. Isolated systolic hypertension in the elderly. JAMA. 1991 Jun 26;265(24):3301-2. No abstract available. PMID 2046114
- [Derived] Chen L, You S, Ee N, Rockwood K, Ward DD, Woodward M, Liu T, Gao Y, Williamson JD, Anderson CS, Harris K, Chen X, Peters R. Impact of Frailty on Antihypertensive Treatment in Older Adults. Hypertension. 2025 Mar;82(3):509-519. doi: 10.1161/HYPERTENSIONAHA.124.24214. Epub 2025 Jan 14. PMID 39807596
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307
- Available data/document: Individual Participant Data Set: SHEP — http://biolincc.nhlbi.nih.gov/studies/shep/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/shep/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/shep/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/shep/